CLINICAL TRIAL: NCT07346716
Title: Medication Concentrations in Human Milk (MedMilk) and Potential Adverse Effects in Breastfed Infants: an Exploratory Clinical Study
Brief Title: Medicines in Breast Milk and Estimated Infant Exposure
Acronym: MedMilk
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jón Þór Trærup Andersen, Professor, PhD,, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-23062687
Record Dates: First submitted 2025-12-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Medication Safety; Lactation; Drug Exposure Via Breast Milk; Pharmacokinetic Parameters
Keywords: breastfeeding; lactation; drug transfer into breast milk; medication safety
MeSH Terms: conditions — Breast Feeding | interventions — Prescription Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breast milk urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breastfeeding women on medication
  Interventions: Drug: Prescription Drugs

INTERVENTIONS:
Drug: Prescription Drugs — Exposure to prescription medicines taken by breastfeeding women during routine treatment. The study does not assign medications but observes drug transfer into human milk from exposures occurring as part of usual care.

SUMMARY:
The MedMilk (Medication concentrations in human Milk) study investigates how selected medicines taken by breastfeeding women are transferred into human milk and whether this may affect the breastfed child. The study includes breastfeeding women who are already using prescription or over-the-counter medicines as part of their usual care. Participants provide samples of breast milk and urine and complete a questionnaire about maternal and infant health. The collected data will be used to quantify medicine concentrations in milk and estimate the relative infant dose. The study aims to contribute new data to support safer prescribing and more informed counselling during breastfeeding

DETAILED DESCRIPTION:
The MedMilk (Medication concentrations in human Milk) study is a prospective, exploratory clinical study coordinated by the Department of Clinical Pharmacology, Bispebjerg and Frederiksberg Hospital, Denmark. The study is observational in nature and involves no experimental drug administration. Participants are breastfeeding women using medicines as part of their routine treatment.

Each participant will provide four small breast milk samples (1-20 mL each) collected at different time points in relation to maternal drug intake, one urine sample, and questionnaire data on maternal and infant health, breastfeeding patterns, and any infant symptoms potentially related to drug exposure. Samples are stored at -80 °C in a dedicated research biobank until analysis.

Drug concentrations in milk and urine will primarily be quantified using solid Phase Extraction coupled with UPLC-MS/MS. Data will be analyzed descriptively, and relative infant doses (RID) will be calculated. For drugs with sufficient sampling density.

Results will add to the limited body of systematic data on drug transfer into human milk and help inform clinical decision-making regarding medication use during breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women aged ≥18 years
* Current use of one or more prescription or over-the-counter (classified within the ATC system) drugs
* Able and willing to provide written informed consent

Exclusion Criteria:

* Current pregnancy during sample collection
* Known and clinically significant pharmacokinetic drug-drug interactions at the time of sampling

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be lactating women recruited through obstetric, neonatal, and psychiatric departments, public health visiting nurses, and counselling services across Denmark. Recruitment will be coordinated by the Department of Clinical Pharmacology, Bispebjerg and Frederiksberg Hospital, Copenhagen. The study primarily targets women using prescription and over-the-counter medicines during breastfeeding and aims to represent real-world exposure patterns across all Danish regions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Drug concentrations in human milk | Within one dosing interval
  Quantification of drug concentrations in human milk, expressed in micrograms per millilitre (µg/mL). Milk samples are collected before and after the maternal dose within one dosing interval.

SECONDARY OUTCOMES:
Relative Infant Dose (RID) | Within one dosing interval
  Estimation of infant drug exposure, expressed as the relative infant dose (% of maternal weight-adjusted dose).
Maternal-reported infant adverse effects | At the time of inclusion. Montly follow-up for three months.
  Maternal questionnaire on infant symptoms potentially related to drug exposure via breastfeeding.

OTHER OUTCOMES:
Simulated infant plasma levels | During one dosing interval
  We will estimate the infant plasma level of the specific drug expressed as microgram pr. millilitre μg/ml based on pharmacokinetic modelling of infant, and drug characteristics and drug concentrations in milk samples.
Simulated Area Under the Curve (AUC) | During one dosing interval
  We will estimate the 95th percentile of the pediatric Area Under the Curve (AUC) (μg x h/mL) based on pharmacokinetic modelling of infant, and drug characteristics and drug concentrations in milk samples.
Biobank establishment | Within one dosing interval
  Milk and urine samples stored for future pharmacokinetic analyses and secondary research

CONTACTS AND LOCATIONS:
Overall Officials: Jon Traerup Andersen, Professor, MD, PhD, Principal Investigator — Department of Clinical Pharmacology, Bispbjeg and Frederiksberg Hospital
Locations (3):
- Denmark (3):
  - Department of Clinical Pharmacology, Copenhagen
  - Mental health services, Capital Region of Denmark, Copenhagen
  - Department of Obstetrics and Gynecology, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol, SAP and ICF after protocol publication. Analytical code and summary results after completion of data collection and analyses.
Access Criteria: Requests for data access can be directed to the principal investigator. Data sharing will require relevant approvals under Danish GDPR.